CLINICAL TRIAL: NCT02473172
Title: Impact of Pressure Support Ventilation (PSV) Versus Neurally Adjusted Ventilatory Assist (NAVA) Diaphragm Efficiency
Brief Title: Impact of the Assisted Ventilation Mode on Diaphragm Efficiency in Critically Ill Patients
Acronym: NAVA_PSV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Salvatore Grasso, Associate Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAVA_PSV
Record Dates: First submitted 2015-06-08; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Respiratory Insufficiency
Keywords: Weaning from mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure Support Ventilation (Experimental): Assisted mechanical ventilation
  Interventions: Device: Pressure Support ventilation
- Neurally Adjusted Ventilatory Assist (Experimental): Assisted mechanical ventilation
  Interventions: Device: Neurally Adjusted Ventilatory Assist

INTERVENTIONS:
Device: Pressure Support ventilation — Assisted mechanical ventilation
  Arms: Pressure Support Ventilation
Device: Neurally Adjusted Ventilatory Assist — Assisted mechanical ventilation
  Arms: Neurally Adjusted Ventilatory Assist

SUMMARY:
This study evaluates the impact of the assisted mode of mechanical ventilation on diaphragm efficiency in mechanically ventilated critically ill patients. Participants will be randomized to the neurally adjusted ventilatory assist (NAVA) mode or to the pressure support ventilation (PSV) mode.

DETAILED DESCRIPTION:
During mechanical ventilation the ventilator applies positive pressure to the respiratory system. Often in the acute phase of critical illness patients are ventilated in the control mode (CMV), where the patient is completely passive. This quickly (within 48 hours) has been shown to induce diaphragm atrophy and dysfunction (Levine et al New England Journal of Medicine, 200; 358:1327-35). To preserve diaphragm function, guidelines suggest to shift as soon as possible to the assisted mode (the ventilator applies positive pressure to assist spontaneous inspiratory effort). The synchrony between patient and ventilator is critical in this context. PSV is the classical assisted mode and applies a constant pressure whatever the patient effort. NAVA is a newer mode based on the diaphragm electrical activity (EAdi) measurement. It assist patient effort proportionally to the EAdi and hence to patient's effort. The investigator hypothesis is that NAVA would improve diaphragm efficiency more efficiently than PSV.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* oro-tracheally or naso-tracheally intubate
* had been ventilated for acute respiratory failure in control mechanical ventilation for at least 72 hours consecutively
* candidate to assisted ventilation
* Hemodynamically stable without vasopressor or inotropes (excluding a dobutamine and dopamine infusion lower than 5 gamma/Kg/min and a 3 gamma /Kg/min, respectively
* normothermia

Exclusion Criteria:

* Neurological or neuromuscular pathologies
* phrenic nerve dysfunction
* contraindications to the insertion of a nasogastric tube (for example recent upper gastrointestinal surgery, esophageal varices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Diaphragm neuro-ventilatory efficiency (NVE) | 48 hours
  Diaphragm neuro-ventilatory efficiency (NVE) to convert the electrical diaphragm activity (EAdi) into volume. NVE is impaired by controlled mechanical ventilation (CMV) and the assisted mode should serve to restore it. All the studied patents were ventilated for more than 48 hours in CMV, a period shown to be sufficient to induce diaphragm atrophy and therefore depress NVE. NVE is measured by the ratio between tidal volume (VT) and the EAdi peak (NVEpeak) or by the ratio between VT and the are under the EAdi signal. EAdi is obtained by the EAdi catheter, a nasogastric catheter equipped with electrodes (Maquet Critical Care, Solna, Sweden). EAdi is measured in microVolt. The Servo i ventilator (Maquet Critical Care, Solna Sweden) is equipped with a module able to amplify and show on a screen the EAdi trace and the corresponding value. Both the Servo i ventilator and the EAdi catheter are approved for clinical use.

SECONDARY OUTCOMES:
Diaphragm neuro-mechanical efficiency (NME) | 48 hours
  Diaphragm neuro-mechanical efficiency (NME) to convert the electrical diaphragm activity (EAdi) into negative pressure is impaired by controlled mechanical ventilation (CMV). The assisted mode should serve to restore it. All the studied patents are ventilated for more than 48 hours in CMV, a period shown to be sufficient to induce diaphragm atrophy and hence depress NME.
  NME is measured by simultaneously recording EAdi and airway opening pressure during an end-expiratory airway opening occlusion and expressed in centimeters of waters (cmH2O)/microVolt.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Grasso, Prof, Principal Investigator — University of Bari
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico, Bari, Italy

REFERENCES:
- [Derived] Di Mussi R, Spadaro S, Mirabella L, Volta CA, Serio G, Staffieri F, Dambrosio M, Cinnella G, Bruno F, Grasso S. Impact of prolonged assisted ventilation on diaphragmatic efficiency: NAVA versus PSV. Crit Care. 2016 Jan 5;20:1. doi: 10.1186/s13054-015-1178-0. PMID 26728475